CLINICAL TRIAL: NCT01038869
Title: Efficacy and Safety of Finacea in the Treatment of Post-Inflammatory Hyperpigmentation and Acne Vulgaris
Brief Title: Efficacy and Safety Study of Finacea to Treat Acne Vulgaris and Post-Inflammatory Hyperpigmentation (PIH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Principal Investigator, Derm Research, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIN0901
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Acne Vulgaris; Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation | interventions — azelaic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azelaic acid 15% (Finacea) (Experimental): Open label pilot study, Topical gel to be appiled twice daily for 16 weeks
  Interventions: Drug: Azelaic acid

INTERVENTIONS:
Drug: Azelaic acid — Apply sparingly to the face twice a day (morning and night). Massage gently into the skin until vanishing. Approximately 0.5g (2.5cm strip) is sufficient for the entire facial area.
  Other Names: Finacea

SUMMARY:
Residual post-inflammatory hyperpigmentation (PIH)from acne is disturbing to individuals with skin of color. Finacea has been anecdotally known to be beneficial in resolving PIH related to acne vulgaris. However, it has not been clinically tested for this purpose. The current study will investigate the efficacy and safety of Finacea in the treatment of acne vulgaris and PIH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 12 years of age
* Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline
* Fitzpatrick skin type IV to VI
* Acne IGA (Investigator Global Assessment) score of 2 or 3
* Inflammatory lesions of 15-60 (with no more than 2 nodules)
* Non-inflammatory lesions of 20-100
* Post Inflammatory Hyperpigmentation Investigator Global Assessment (PIH IGA) score of 3,4 or 5
* Able to understand the requirements of the study and sign Informed Consent/HIPAA forms. Subjects under the legal age of consent must have the written informed consent of a parent or legal guardian

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding or who are of childbearing potential and not practicing a reliable method of birth control
* Allergy or sensitivity to any component of the test medication
* Subjects who have not complied with the wash out periods for prohibited medications
* Medical condition that contraindicates participation
* Skin disease/disorder that might interfere with the diagnosis of acne vulgaris or PIH
* Evidence of recent alcohol or drug abuse
* History of poor cooperation, non-compliance or unreliability
* Exposure to an investigational drug study within 30 day of Baseline visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from private office population.
Groups:
- Finacea: Open label pilot study. All subjects were given Azelaic acid 15% to be used topically, twice daily.
Period: Overall Study
Arm/Group | Finacea
Started | 20
Completed | 13
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Groups:
- Finacea: Open label pilot study
Arm/Group | Finacea
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement in Acne IGA (Investigator Global Assessment)
Description: IGA Assessments at each visit (baseline and follow up) based on a 6 point scale (0= clear through 5 = very severe). Improvement is defined as at least a 1 point improvement.
Time Frame: Baseline to 16 weeks
Population: Per protocol
Measure: Number; unit: percentage of participants
Groups:
- Azelaic Acid 15% Open Label: Assessments of IGA
Arm/Group | Azelaic Acid 15% Open Label
Number analyzed (Participants) | 20
percentage of participants | 92

2. Secondary Outcome: Percentage of Participants With Improvement in the IGA of Post Inflammatory Hyperpigmentation(PIH)
Description: IGA for PIH assessed on a 7 point scale (0= clear through 6 = severe) with at least a two point improvement
Time Frame: Baseline to16 weeks
Population: per protocol
Measure: Number; unit: percentage of participants
Groups:
- Azelaic Acis 15% Open Label: Assessments of PIH IGA
Arm/Group | Azelaic Acis 15% Open Label
Number analyzed (Participants) | 20
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With an Improvement in Post Inflammatory Hyperpigmentation (PIH) % Distribution
Description: The % distribution of PIH, evaluated on a scale of 0 = no PIH through 6 = greater than 50%
Time Frame: Baseline to 16 weeks
Population: per protocol
Measure: Number; unit: percentage of participants
Arm/Group | Azelaic Acid 15%
Number analyzed (Participants) | 20
percentage of participants
  2 grade improvement | 92
  1 grade improvement | 100

4. Secondary Outcome: Percentage Change in Total Lesion Counts
Description: Total lesions including inflammatory lesions (papules, pustules, nodules) and non-inflammatory lesions (open and closed comedones).
Time Frame: Baseline to 16 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: percentage of total lesion count
Groups:
- Azelaic Acid 15%: lesion counts
Arm/Group | Azelaic Acid 15%
Number analyzed (Participants) | 20
percentage of total lesion count | -92.4 (10.4)

5. Secondary Outcome: Tolerability Assessments as Measured by the Number of Participants With Side Effects
Description: Tolerability parameters assesssed by the presence and degree of peeling, erythema, dryness, oiliness, burning and pruritus
Time Frame: 16 weeks
Population: per protocol
Measure: Number; unit: participants
Groups:
- Azelaic Acid 15%: tolerability assessments
Arm/Group | Azelaic Acid 15%
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Arm/Group | Finacea
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This is an open-label study with a small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes